CLINICAL TRIAL: NCT02513602
Title: Peri-Implant Bone Assessment in Transplanted Patients: A Case Control Study
Brief Title: Osseointegrated Dental Implants in Kidney Transplanted Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Trieste (Other)
Responsible Party: Principal Investigator, prof. Roberto Di Lenarda, Professor, University of Trieste
Other Study IDs: ITR
Record Dates: First submitted 2015-07-20; First posted 2015-07-31 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Tooth Loss; Disorder Related to Renal Transplantation
Keywords: implantology; kidney; renal disease; edentulism; tooth loss
MeSH Terms: conditions — Tooth Loss; Kidney Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — bone specimen harvested during implant site preparation in order to obtain usefull samples for hystomorphometrical analysis
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- TEST group (kidney transplanted): Kidney transplanted patients, passed through dialysis phase presenting a mandibular edentulism. It will be scheduled one or two dental implants to be inserted in mandible.
  This group will be subjected to a dental implant insertion procedure.
  Interventions: Procedure: Dental implant insertion
- CONTROL group (healthy patients): Healthy patients, with an inserted mandibular implant, retrospectively enrolled with a preoperative cbct scan.

INTERVENTIONS:
Procedure: Dental implant insertion — Dental implant insertion will be carry out in the mandible of the patients enrolled, through a surgical template in order to repeat the same position of the simulating implant insertion. After a trephine bur passage, the final two or three twist-drills will be used to realize the implant socket. After implant positioning, a cover screw will be tightened and the mucosa sutured above.
  Groups: TEST group (kidney transplanted)

SUMMARY:
The evaluation of the bone, using several techniques and on several aspects will be the purpose to study the possible impact of the kidney transplant (and, extensively, the pre-transplant dialysis, the organ replacement and the immunosuppressive therapy) could have on the bone metabolism and on the density of the bone where the implants are placed. The assessment on the bone density only in a retrospectively selected population that underwent the same surgical procedure will help the comparison of the data to get a satisfactory conclusion. The evaluation of other clinical and instrumental parameters in the test group makes the kidney-transplant patients bone quality clear, and will consequently demonstrate if implants are a feasible therapy for these patients.

DETAILED DESCRIPTION:
The primary purpose of this study is the evaluation of the effects of the kidney transplant on the periimplant bone density by the comparison with the density of healthy patients. The secondary purpose is obtaining clinical, histological and radiographic data to evaluate the effect of systemic conditions and its rebound on the insertion of fixtures.

Evaluation criteria

1. Control group: evaluation of the periimplant bone density (1 mm) next to the implant virtually planned using the CT editing software on the cone beam CT acquired in a retrospective sample of patients already treated with the insertion of a fixture in the molar or premolar edentulous site
2. Test group: periodontal evaluation with plaque index, bleeding on probing index and probing 1 month before operation.
3. Test group: evaluation of periimplant bone density (1 mm) in the fixture virtual-projected zone (the implant will be inserted there) with the CT acquisition and editing software.
4. Test group: evaluation of the implant stability after their insertion (primary stability) using the Resonance Frequence Analysis. ISQ (Implant Stability Quotient) value is expressed in 4 numbers (mesial, distal, buccal, lingual), average values of three measures acquired in each side.
5. Test group: evaluation of the implant stability immediately after the insertion calculating the insertional torque value (ITV) with an implant motor.
6. Test group: evaluation of the periimplant bone using an endoral periapical radiograph with Rinn device immediately after the operation.
7. Test group: histomorphological examination of the bone core sample made by a trephine resulted from the implant site preparation

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: single or partial mandibular molar-premolar edentulism that requires up to 2 fixtures
* Good systemic compensation of the kidney transplant (≤ ASA American Society of Anesthesiologists score 3) with at least 1 year of previous hemodialysis or peritoneal dialysis and in actual immunosuppressive therapy
* Be older than 18 years
* The patient must be able to understand the meaning of the study and accept to undergo periodical follow-up controls.
* The patient must be able to understand and practice all the oral hygiene procedures demanded by the experimenter
* Signature of the informed consent form

and for control

* Diagnosis: single or partial mandibular molar-premolar edentulism that requires up to 2 fixtures
* Having a pre-operatory cone beam CT available
* Age older than 18 years
* Signature of the authorization to use and process personal details at the acceptance of every sort of treatment in the Company Hospital of Trieste.

Exclusion Criteria:

* Post extraction implant (before 3 months from the extraction)
* Be less than 18 years old
* Smoking more than 10 cigarettes/day
* Plaque index more than 25
* Bleeding on probe index more than 25
* Clear allergy or intolerance against the products used in the study
* Patients that require reconstructive bone surgery before the fixtures placement (gbr and bone grafting)

and for control group

* Patients that require reconstructive bone surgery before the fixtures placement (gbr and bone grafting)
* Pathologies and pharmacological therapies that interfere with bone (for instance osteoporosis, osteomalacia, malnutrition, Paget's disease, corticosteroid therapy, bisphosphonate therapy, head and neck radiotherapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The minimal number of the participants of this study is 26 per group: this results from the measure of a 0,8 effect size. If the effect size is less than 1 (minimal value), it represents the situation where the medium difference of standard deviations of the variable "bone density" is equivalent to the difference of the value between the two groups of the study.
  Subject of test group will be enrolled an a kidney transplanted patients, while Subjects of control group will be enrolled retrospectively in healthy patients
Sampling Method: Probability Sample
Enrollment: 26 (Estimated)
Dates: Start 2014-05; Primary Completion 2020-05 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Bone density measured in Grey Value | seven days after cone beam computed tomography
  bone density will be assessed on the cone beam CT scans with the virtual implant positioning before surgery (for the test group) and postoperatively (retrospectively assessed) for the control group. Grey Value will be assessed in the area of 1 mm around the shape of the implants.

SECONDARY OUTCOMES:
Insertional torque value | during implant placement
  Only for the test group the Insertional torque value will be assessed during surgery.
Histomorphometric analysis | within 20 days after implant placement
  Only for the test group the microscopic analysis will be performed on the specimen harvested during surgery (via trephine bur, preparing the implant site)

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Di Lenarda, DDS, MSc, Study Director — University of Trieste Medical School, Department of Odontology and Stomatology
Locations (1):
- University Hospital Company, "Ospadale Maggiore", Trieste, TS, Italy

REFERENCES:
- [Background] Arisan V, Karabuda ZC, Avsever H, Ozdemir T. Conventional multi-slice computed tomography (CT) and cone-beam CT (CBCT) for computer-assisted implant placement. Part I: relationship of radiographic gray density and implant stability. Clin Implant Dent Relat Res. 2013 Dec;15(6):893-906. doi: 10.1111/j.1708-8208.2011.00436.x. Epub 2012 Jan 17. PMID 22251553
- [Background] Cassetta M, Stefanelli LV, Di Carlo S, Pompa G, Barbato E. The accuracy of CBCT in measuring jaws bone density. Eur Rev Med Pharmacol Sci. 2012 Oct;16(10):1425-9. PMID 23104660
- [Background] Zou H, Zhao X, Sun N, Zhang S, Sato T, Yu H, Chen Q, Weber HP, Dard M, Yuan Q, Lanske B. Effect of chronic kidney disease on the healing of titanium implants. Bone. 2013 Oct;56(2):410-5. doi: 10.1016/j.bone.2013.07.014. Epub 2013 Jul 19. PMID 23876979